CLINICAL TRIAL: NCT03144531
Title: Sleep Intervention for Kids and Parents (SKIP): A Self-Management Pilot Study
Brief Title: Sleep Intervention for Kids and Parents: A Self-Management Pilot Study
Acronym: SKIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jennifer Sonney, Assistant Professor, Family and Child Nursing, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001834; P30NR016585-01 (NIH)
Record Dates: First submitted 2017-05-01; First posted 2017-05-08 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Sleep Disturbance; Asthma
Keywords: School-age child
MeSH Terms: conditions — Parasomnias; Asthma

STUDY DESIGN:
Intervention Model Description: Dyadic intervention for school-age children and a parent
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKIP Intervention (Experimental)
  Interventions: Behavioral: Sleep Intervention for Kids and Parents (SKIP)

INTERVENTIONS:
Behavioral: Sleep Intervention for Kids and Parents (SKIP) — Dyadic approach using self-efficacy theory to set goals, anticipate barriers, problem solve

SUMMARY:
Behavioral intervention for 6-11 year children with persistent asthma and sleep disturbance and a parent with sleep disturbance.

ELIGIBILITY:
Inclusion Criteria (child):

* Children 6-11 years
* Child diagnosis of asthma with prescription for daily medication
* Able to understand English (child)
* Sleep disturbance per CSHQ (child >= 41) and/or < 9 hours of sleep per night

Exclusion Criteria (child)

* Parent reported diagnosis of traumatic brain injury, developmental delay, autism spectrum disorder, attention deficit hyperactivity disorder (ADHD), obstructive sleep apnea, cancer
* Positive sleep related breathing disorder screening (obstructive sleep apnea screening)

Inclusion Criteria (parent)

* 18 years or older
* Able to understand and read English
* Lives with child 50% of time or more
* Is child's legal guardian
* Has reliable access to internet
* >/= 5 on Pittsburgh Sleep Quality Index or <7 hours overnight reported sleep

Exclusion Criteria (parent)

* Diagnosed obstructive sleep apnea or sleep disordered breathing
* Is a nightshift worker
* Uses sleep medication

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Total sleep time | 3 months post intervention (x 10 days of measurement)
  Actigraphy
Sleep efficiency | 3 months post intervention (x 10 days of measurement)
  Actigraphy
Bedtime Consistency | 3 months post intervention (x 10 days of measurement)
  Actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sonney, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Nursing, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sonney JT, Thompson HJ, Landis CA, Pike KC, Chen ML, Garrison MM, Ward TM. Sleep intervention for children with asthma and their parents (SKIP Study): a novel web-based shared management pilot study. J Clin Sleep Med. 2020 Jun 15;16(6):925-936. doi: 10.5664/jcsm.8374. PMID 32056537